CLINICAL TRIAL: NCT05730868
Title: Effect of Exercise Among Turtle Neck Syndrome in Pakistani Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Karachi (Other)
Responsible Party: Principal Investigator, Khadija Tul Kubra, PT, Assistant Professor, University of Karachi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KTKYasin
Record Dates: First submitted 2023-01-20; First posted 2023-02-16 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Neck Pain
Keywords: text neck syndrome; neck pain; Turtle neck syndrome; tissue hardness; pain pressure threshold
MeSH Terms: conditions — Neck Pain | interventions — Myofascial Release Therapy

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- group 1 myofascial release (Experimental): soft tissue release technique to release tension from muscles which relieves pain and increase range of motion
  Interventions: Procedure: myofascial release
- group 2 muscle energy technique (Experimental): soft tissue release technique to release tension from muscles which relieves pain and increase range of motion
  Interventions: Procedure: muscle energy technique
- group 3 MFR & MET (Experimental): combination of two soft tissue release techniques to release tension from muscles which relieves pain and increase range of motion
  Interventions: Procedure: MFR & MET
- group 4 conventional therapy (Experimental): combination of traditional techniques to relieve pain and spasm
  Interventions: Procedure: conventional therapy

INTERVENTIONS:
Procedure: myofascial release — Soft tissue release will be performed on the trapezius, sub occipital and sternocleidomastoid muscles. The visual analog scale will be used to check pain intensity. Algometer will be used to check the pain pressure threshold and tissue hardness. neck disability index will be used to check neck disability
  Arms: group 1 myofascial release
Procedure: muscle energy technique — Muscle energy Technique will be performed on the trapezius, sub occipital and sternocleidomastoid muscles. The visual analog scale will be used to check pain intensity. Algometer will be used to check the pain pressure threshold and tissue hardness. neck disability index will be used to check neck disability
  Arms: group 2 muscle energy technique
Procedure: MFR & MET — combination of myofascial release and muscle energy technique will be performed on the trapezius, suboccipital and sternocleidomastoid muscles. The visual analog scale will be used to check pain intensity. Algometer will be used to check the pain pressure threshold and tissue hardness. neck disability index will be used to check neck disability
  Arms: group 3 MFR & MET
Procedure: conventional therapy — traditional physical therapy devices are used to relieve pain and spam. this will include a hot pack, ultrasound, and TENS (Transcutaneous electrical nerve stimulation)
  Arms: group 4 conventional therapy

SUMMARY:
Turtle neck also known as Text neck or anterior head syndrome is an overuse syndrome which occurs due to repetitive stress to neck, either by hanging it down or forward using phone or electronic devices. Typical signs and symptoms include pain and stiffness in the neck, shoulder pain and increase curvature of spine. It is becoming a global burden as people of almost all ages are getting affected.

The objective of the study is to find out theEffect of Exercise among Turtle Neck Syndrome in Pakistani Population. A total of 100 participants will be included in the study having both males and females. The pain pattern will be assessed by Visual Analog Scale and Posture Grid Assessment tool will be used to assess posture before and after the treatment session.

The study will be divided into three main sections or groups. One group will be treated by myofascial release only while other group will be treated by muscle energy technique for the management of turtle neck syndrome. Third group will receive both MFP and MET exercise. People having neck pain and those who will be willing to participate will be included in the study.

DETAILED DESCRIPTION:
The participants will be divided into four groups namely group A, B, C and D. Initially all the participants will be assessed by posture grid assessment tool to check their postural deviations. People meeting the inclusion criteria will be recruited. Group A will receive Muscle Energy Technique (MET) exercise, Group B will receive Myofascial release (MFP) therapy, Group C will receive both MFP and MET and group D will receive conventional treatment. Pre and post Visual analog scale (VAS) will be used to check pain scale and posture grid assessment tool to check postural angles .Pre-assessment will be done on day one and post at the last day of session. The total duration of treatment will be four weeks.

Consent will be taken from the patients. Only those patients meeting the inclusion criteria and screening questions will included in the study and those who will be willing to participate.

ELIGIBILITY:
Inclusion Criteria:

* both males and females will be included
* patients having non specific neck pain
* usage of mobile more than six hours
* patients willing to participate

Exclusion Criteria:

* pregnant females
* patients having cervical disc bulge or herniation disoriented patients
* patients not willing to participate
* patients having any deformity

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
visual analog scale | 2 years
  For pain intensity visual analog scale will be used. a patient oriented scale ranging from 0-10. 0 means no pain, 1-3 means mild pain, 4-6 means moderate pain and 7-10 means severe pain.
Neck disability Index | 2 years
  to check disability, Neck disability Index will be used. It's a ten section questionnaire. Each item has scoring of 0-5. For each section the total possible score is 5.
  Points are summed to a total score. 0-4points (0-8%) no disability, 5-14points ( 10 - 28%) mild disability, 15-24points (30-48% ) moderate disability, 25-34points (50- 64%) severe disability, 35-50points (70-100%) complete disability
The tissue hardness assessed by Algometer measured in Newtons | 2 years
  For tissue hardness, Algometer will be used. It's a device that calculates the hardness when given pressure against the stimuli. The value is measured in Newtons.
Pain pressure threshold assessed by Algometer measured in Newtons | 2 years
  For Pain pressure threshold, Algometer will be used. It's a device that calculates the pain pressure threshold when given pressure against the stimuli. The value is measured in Newtons.

CONTACTS AND LOCATIONS:
Overall Officials: Khadija Tul Kubra, M.phil, Principal Investigator — University of Karachi
Locations (1):
- Khadija, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
no their is no plan to share IPD

REFERENCES:
- [Background] Ajimsha MS, Al-Mudahka NR, Al-Madzhar JA. Effectiveness of myofascial release: systematic review of randomized controlled trials. J Bodyw Mov Ther. 2015 Jan;19(1):102-12. doi: 10.1016/j.jbmt.2014.06.001. Epub 2014 Jun 13. PMID 25603749
- [Background] Phadke A, Bedekar N, Shyam A, Sancheti P. Effect of muscle energy technique and static stretching on pain and functional disability in patients with mechanical neck pain: A randomized controlled trial. Hong Kong Physiother J. 2016 Apr 14;35:5-11. doi: 10.1016/j.hkpj.2015.12.002. eCollection 2016 Dec. PMID 30931028
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/30931028/